CLINICAL TRIAL: NCT03476759
Title: Laparoscopic Tubal Adhesiolysis Versus IVF-ICSI in Cases of Post Caesarean Section Adhesions, Which is the Best?
Brief Title: Laparoscopic Tubal Adhesiolysis Versus IVF-ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tanta University
Record Dates: First submitted 2018-03-18; First posted 2018-03-26 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Tubal Factor Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tubal adhesiolysis (Active Comparator): laparoscopic tubal adhesiolysis and\or tuboplasty
  Interventions: Procedure: Tubal adhesiolysis
- IVF/ICSI (Active Comparator): These patients will undergo IVF/ICSI
  Interventions: Drug: IVF/ICSI

INTERVENTIONS:
Procedure: Tubal adhesiolysis — 125 patients will undergo tubal adhesiolysis or tuboplasty
  Arms: Tubal adhesiolysis
Drug: IVF/ICSI — 125 patients will undergo IVF-ICSI procedures.
  Arms: IVF/ICSI

SUMMARY:
2groups with peritoneal adhesions after cesarean delivery will be allocated to either laparoscopic tubal adhesiolysis or to IVF/ICSI

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at Tanta university hospitals in fertility and MIS units. Two hundred and fifty 2ry infertility patients with confirmed post C.S adhesions will be included in the study and those patients will be divided randomly in two groups:

Group A:

125 patients will be undergoing laparoscopic tubal adhesiolysis and\or tuboplasty then a widow of 12 months post operatively is given for natural conception.

Group B:

125 patients will undergo IVF-ICSI procedures. The primary outcome measure of the study will be the rate of clinical pregnancy.

Inclusion criteria:

* patient's age not exceeding 35 years old
* confirmed post caesarean section tubal adhesions (by diagnostic laparoscopy report or video CDs) as a solitary cause of their 2ry infertility.

Exclusion criteria:

* patient's age >35 years
* other causes of infertility as male factor contribution, any ovulatory or endocrinological disorder,
* diagnosed any degree of endometriosis
* patients with history of recurrent pregnancy loss.
* couples with prolonged sexual abstinence for any reason Detailed explanation of the aims, procedures, steps and nature of the study for the participants will be done and a written consent will be signed by each patient before inclusion.

After allocation laparoscopic tubal adhesions will be dissected and normal anatomy and function will be restored. In the other group IVF/ICSI will be commenced The follow up with both groups will extend to 1year or till pregnancy is aggrieved The outcomes of the study were pregnancy rates and affordability

ELIGIBILITY:
Inclusion Criteria:

* age not exceeding 35 years old with confirmed post caesarean section tubal adhesions (by diagnostic laparoscopy report or video CDs) as a solitary cause of their 2ry infertility.

Exclusion Criteria:

* patient's age >35 years, male factor contribution, any ovulatory or endocrinological disorder, diagnosed any degree of endometriosis and patients with history of recurrent pregnancy loss. Couples with prolonged sexual abstinence for any reason will be excluded from participation in the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females only
Enrollment: 300 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | After 1year
  The number of pregnant women in both groups

OTHER OUTCOMES:
Affordability | Within 1year
  Costs of each maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Dawood, MD, Principal Investigator — Lecturer at Tanta University
Locations (1):
- Ayman Shehata Dawood, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
yes